CLINICAL TRIAL: NCT03225118
Title: Comprehensive Evaluation of the Impact of a Short-Term Analytical Treatment Interruption and Re-Initiation of Antiretroviral Therapy on Immunologic and Virologic Parameters in HIV-Infected Individuals
Brief Title: Impact of a Short-Term Analytical Treatment Interruption and Re-Initiation of Antiretroviral Therapy on Immunologic and Virologic Parameters in HIV-Infected Individuals
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170106; 17-I-0106
Record Dates: First submitted 2017-07-20; First posted 2017-07-21 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: HIV
Keywords: Rebound; Reinitiation; ART; Reservoirs; Immune Exhaustion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV/ATI: HIV-infected Adults (age 18-65 years) on ART with suppressed viremia willing to interrupt treatment and then restart once criteria is met.

SUMMARY:
Background:

The immune system helps the body fight off disease. Most people infected with HIV cannot control the infection and need daily medicine. Combination antiretroviral therapy (cART) are drugs taken to prevent HIV infection from damaging the immune system. Researchers want to study why some people develop resistance to the drugs or have permanent side effects.

Objective:

To study the impact of a short-term treatment stop on HIV that persists even while taking cART.

Eligibility:

Adults 18-65 years old with HIV who are being treated with cART

Design:

* Participants will first be screened with a physical exam and medical history. They may have a chest x-ray. They will have heart, blood, and urine tests.
* At the baseline visit, participants will repeat the screening tests except the x-ray. They will get counseling about HIV and risk behavior.
* Participants will have leukapheresis. Blood will be removed through a needle in one arm. A machine will separate white blood cells from the rest of the blood. The remainder of the blood will be returned to the body by a different needle.
* Participants will stop their current treatment on day 0. They will visit the clinic each week until they meet the criteria to restart cART. These visits will have the same procedures as the baseline visit.
* Before restarting cART, most participants will have leukapheresis.
* After restart, participants will be seen weekly for 4 weeks and then monthly for about 11 months. Participants will have blood drawn, physical exam, and medical history. They will have leukapheresis 2 more times over 1 year.

DETAILED DESCRIPTION:
While antiretroviral therapy (ART) has improved the clinical outcome for HIV-infected individuals, persistence of viral reservoirs in the peripheral blood and lymphoid tissues remains a hurdle to the eradication of virus. The vast majority of HIV-infected individuals treated with ART experience plasma viral rebound within weeks of cessation of therapy. Considering that current research regarding treatment has been heavily focused on developing strategies aimed at achieving sustained virologic remission in the absence of ART, it is of crucial importance to investigate the impact of short-term treatment interruption and re-initiation of ART on transcriptional, immunologic, and virologic parameters in HIV-infected individuals. Currently, much of our knowledge regarding the mechanism of viral rebound is based on investigations using structured treatment interruptions in supervised clinical settings dating back to 1999. Subsequent studies, performed primarily in chronically infected patients to minimize treatment exposure and toxicity, revealed poor outcomes in terms of viral rebound, clinical events and mortality 3-11 leading to the abandonment of this genre of investigation. However, various aspects have been identified as potential contributors to the observed negative outcomes including outmoded ART regimens, infrequent post-interruption monitoring, and repeated cycles of prolonged analytical treatment interruption (ATI). While long-term ATI was found to be associated with a decrease in CD4+ T cells, persistent plasma viremia, and an increased risk of opportunistic infections, it is unclear whether short term ATI elicits similar immunologic and virologic consequences in those receiving modern and efficacious ART. Furthermore, the mechanism, kinetics, degree, as well as immunologic and virologic predictors, of plasma viral rebound in patients receiving contemporary antiretroviral drug regimens after cessation of ART have not been explicitly investigated. Nor has the impact of persistent HIV reservoir size been fully correlated to the dynamics of plasma viral rebound in patients receiving modern drug regimens. As we develop clinical trials aimed at therapeutic and curative interventions, an integral component in design will require an ATI phase. Characterizing the corollaries of brief treatment cessation and re-initiation of ART on the dynamics of immunologic parameters and HIV reservoirs will provide valuable information for the design of future trials essential to our interpretation of the results as well as to ensuring the safest environment for the patients. We propose to examine the effect of ATI on plasma viral rebound, changes in immunologic parameters and the dynamics of viral reservoirs in HIV-infected individuals receiving state-of-the-art antiretroviral drug regimens following discontinuation and reinitiation of therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age, 18-65 years
* Documented HIV-1 infection and clinically stable
* In general good health, with an identified primary health care provider for medical management of HIV infection and willing to maintain a relationship with a primary health care provider for medical management of HIV infection while participating in the study
* CD4+ T cell count greater than 450 cells/mm^3 at screening
* Documentation of continuous ART treatment with suppression of plasma viral level below the limit of detection for greater than or equal to 2 years. Subjects with blips (i.e., detectable viral levels on ART) prior to creening may be included provided they satisfy the following criteria:

  * The blips are less than 400 copies/mL, and
  * Succeeding viral levels return to levels below the limit of detection on subsequent testing
* Willingness to undergo ATI
* Willingness to restart ART once restart criteria are met

Laboratory values within pre-defined limits at screening:

* Absolute neutrophil count greater than 1,000/mm^3
* Hemoglobin (Hgb) levels greater than 10.0 g/dL for men and greater than 9.0 g/dL for women
* Platelet count greater than 150,000/mm^3
* Estimated glomerular filtration rate (eGFR) greater than or equal to 60 mL/min as determined by the NIH Clinical Center (CC) laboratory
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels of less than 2.5 x upper limit normal (ULN)

  * Willingness to have samples stored for future research

EXCLUSION CRITERIA:

* Chronic hepatitis B, as evidenced by a positive test for hepatitis B surface antigen (HBsAg), an isolated positive Hepatitis B core antibody (negative HBsAg and anti-HBV Ab) and/or positive Hepatitis B virus (HBV) DNA.
* Chronic hepatitis C virus (HCV) infection as evidenced by a positive test for HCV RNA. Subjects with a positive test for HCV antibody and a negative test for HCV RNA are eligible.
* Has a history of institution of ART within 12 weeks of being diagnosed with acute or early HIV-1, where acute/early infection is defined by any one of the following:

  * Positive HIV-1 enzyme immunoassay (EIA) with negative/indeterminate HIV-1 western blot that subsequently becomes positive
  * Negative HIV-1 EIA within the past 4 months and HIV-1 RNA levels of greater than 400,000 copies/mL, in the setting of a potential exposure to HIV-1.
  * Negative rapid HIV-1 within one month prior to a positive HIV-1 EIA and HIV-1 western blot
  * Low level HIV antibodies (positive EIA or western blot) with a non-reactive detuned EIA
* Documented nadir CD4+ T cell count less than 200 cells /mm^3

  --Patients with a nadir CD4+ T cell count between 100-200 are not excluded, provided their current CD4+ T cell count has been >450 the past 3 years

  ---Subjects with dips (i.e., transient decreases in their CD4 count) prior to screening may be included provided they satisfy the following criteria:
  * a. The dips are > 350 cells/mL, and
  * b. Succeeding CD4 counts return to levels above 450 cells/mL on subsequent testing
* Any history of AIDS defining opportunistic infections
* Subjects with history of receiving ART consisting of mono or dual drug therapy
* Documented multiclass antiretroviral drug resistance that, in the judgement of the investigator, would pose a risk of virologic failure should additional mutations develop during the study
* Any experimental non-HIV vaccination received within 2 weeks prior to study enrollment and at any time during the study.
* Any licensed or experimental non-HIV vaccination (e.g., hepatitis B, influenza, pneumococcal polysaccharide) received within 2 weeks prior to study enrollment/Day 0
* Receipt of other investigational study agent within 28 days of enrollment/day 0 and at any time during the study
* Any active malignancy that may require systemic chemotherapy or radiation therapy
* Systemic immunosuppressive medications received within 3 months prior to enrollment. The following are not excluded: (1)corticosteroid nasal spray or inhaler; (2) topical corticosteroids for mild, uncomplicated dermatitis; and (3) oral/parenteral corticosteroids administered for non-chronic conditions not expected to recur (length of therapy less than or equal to 10 days, with completion in greater than or equal to 30 days prior to enrollment/day 0)
* History of or other clinical evidence of:

  * Significant or unstable cardiac disease (e.g., angina, congestive heart failure, recent myocardial infarction)
  * Severe illness, malignancy, immunodeficiency other than HIV, active systemic infection other than HIV, or any other condition that, in the opinion of the investigator, would make the subject unsuitable for the study
* Active drug or alcohol abuse or any other pattern of behavior that, in the opinion of the investigator, would interfere with adherence to study requirements
* Both male and female subjects to remain completely abstinent of potentially reproductive sexual intercourse (e.g. due to a committed lifestyle) or to consistently use BOTH a barrier method with a spermicide (male or female condom) AND ALSO one of the below listed methods of birth control:

  * Continuous/daily hormonal methods including oral contraceptive pills, patch, implant/injection, etc.
  * Surgical sterilization of either partner, of sufficient duration to be effective, and NOT known to have failed.
  * Intrauterine device.
* Females of childbearing potential must not be breast-feeding, possibly or actually pregnant, must not have had unprotected intercourse for one month prior to enrollment , and must agree not to become pregnant beginning from enrollment in the study to at least 8 weeks after the end of analytical treatment interruption.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV patients which will be recruited from natural history and training protocols currently enrolling in clinic and the community
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
The time to plasma viral rebound in HIV-infected individuals undergoing analytical treatment interruption. | The outcome will be satisfied when each subject meets restart criteria.

SECONDARY OUTCOMES:
The difference in frequency of HIV infected CD4+ and CD8+ T cells and the respective expression of immune exhaustion markers prior to and following ATI and after re-initiation of ART. | The time points to evaluate the outcome differences will be at baseline, during treatment interruption and after cART is restarted.
  The difference in frequency of HIVinfected CD4+ and CDS+ T cells and the respective expression of immune exhaustion markers prior to and following ATI and after re-initiation of ART.

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Sneller, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Davey RT Jr, Bhat N, Yoder C, Chun TW, Metcalf JA, Dewar R, Natarajan V, Lempicki RA, Adelsberger JW, Miller KD, Kovacs JA, Polis MA, Walker RE, Falloon J, Masur H, Gee D, Baseler M, Dimitrov DS, Fauci AS, Lane HC. HIV-1 and T cell dynamics after interruption of highly active antiretroviral therapy (HAART) in patients with a history of sustained viral suppression. Proc Natl Acad Sci U S A. 1999 Dec 21;96(26):15109-14. doi: 10.1073/pnas.96.26.15109. PMID 10611346
- [Background] Bar KJ, Sneller MC, Harrison LJ, Justement JS, Overton ET, Petrone ME, Salantes DB, Seamon CA, Scheinfeld B, Kwan RW, Learn GH, Proschan MA, Kreider EF, Blazkova J, Bardsley M, Refsland EW, Messer M, Clarridge KE, Tustin NB, Madden PJ, Oden K, O'Dell SJ, Jarocki B, Shiakolas AR, Tressler RL, Doria-Rose NA, Bailer RT, Ledgerwood JE, Capparelli EV, Lynch RM, Graham BS, Moir S, Koup RA, Mascola JR, Hoxie JA, Fauci AS, Tebas P, Chun TW. Effect of HIV Antibody VRC01 on Viral Rebound after Treatment Interruption. N Engl J Med. 2016 Nov 24;375(21):2037-2050. doi: 10.1056/NEJMoa1608243. Epub 2016 Nov 9. PMID 27959728
- [Background] Strategies for Management of Antiretroviral Therapy (SMART) Study Group; El-Sadr WM, Lundgren J, Neaton JD, Gordin F, Abrams D, Arduino RC, Babiker A, Burman W, Clumeck N, Cohen CJ, Cohn D, Cooper D, Darbyshire J, Emery S, Fatkenheuer G, Gazzard B, Grund B, Hoy J, Klingman K, Losso M, Markowitz N, Neuhaus J, Phillips A, Rappoport C. CD4+ count-guided interruption of antiretroviral treatment. N Engl J Med. 2006 Nov 30;355(22):2283-96. doi: 10.1056/NEJMoa062360. PMID 17135583
- [Derived] Sneller MC, Huiting ED, Clarridge KE, Seamon C, Blazkova J, Justement JS, Shi V, Whitehead EJ, Schneck RF, Proschan M, Moir S, Fauci AS, Chun TW. Kinetics of Plasma HIV Rebound in the Era of Modern Antiretroviral Therapy. J Infect Dis. 2020 Oct 13;222(10):1655-1659. doi: 10.1093/infdis/jiaa270. PMID 32443148
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-I-0106.html